CLINICAL TRIAL: NCT05686031
Title: An Evaluation of Operating Room Staff's Awareness of Environmental Sustainability and Medical Waste Management
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, Clinical associated professor, Ankara University
Other Study IDs: I4-165-19
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Environmental-Pollution-Related Condition
Keywords: Environment; Inhalational Anaesthetics; Recycling; Global Warming; Carbon Footprint; Operating Room

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Doctors: Anaesthesiologists
  Interventions: Other: No interventions were done between groups
- Anaesthesia Nurses
  Interventions: Other: No interventions were done between groups

INTERVENTIONS:
Other: No interventions were done between groups — No interventions were done between groups

SUMMARY:
The main goals of this single-centre cross-sectional study were to measure views on the environmental effects of the operating room and identify the main barriers to recycling in the operating room environment as perceived by the staff. Participants responded a questionnaire to measure their opinions and the views.

ELIGIBILITY:
Inclusion Criteria:

* all personel working in operating room

Exclusion Criteria:

* missing data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anaesthesiologists, surgeons, residents, nurses, cleaning staff and medical students from any gender and age group working in Ankara University.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Most reported barriers to recycling | 3 Weeks
Views on the environmental effects of the OR | 3 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- AnkaraU, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no intention and approval to share IPD